CLINICAL TRIAL: NCT04123431
Title: A Prospective UK Multi-Centre Post Market Clinical Follow-up Study of the JRI Orthopaedic ACE Acetabular Cup System
Brief Title: ACE Acetabular Cup UK Multi-centre PMCF Study
Status: Recruiting | Type: Observational
Sponsor: JRI Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: JRI-CS-010
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hip Disease
Keywords: Total Hip Replacement; Patient reported outcome measures; Post Market Clinical Follow-up / Post Market Surveillance
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ACE Acetabular Cup System with XLPE Liner
  Interventions: Device: Total Hip Replacement
- ACE Acetabular Cup System with Ceramic Liner
  Interventions: Device: Total Hip Replacement
- ACE Acetabular Cup System with Dual Mobility Insert
  Interventions: Device: Total Hip Replacement

INTERVENTIONS:
Device: Total Hip Replacement — Primary elective total hip replacement

SUMMARY:
A total hip replacement is one of the most successful and cost-effective surgical procedures in orthopaedics, and involves replacing both the hip ball and socket. Its goal is to provide pain relief, allowing the person to return to a normal lifestyle. JRI Orthopaedics have developed the ACE Acetabular Cup System, which has a H-A.C. coating to promote ossoeintegration of the device within the host bone. To increase the surgeons choice and thus suitability for the patient, there is the option of 3 different socket liners (ceramic, polymer or dual mobility).

To ensure maximum safety and performance of medical devices surveillance of the device should be carried out over the devices lifetime. This study is a 10 year surveillance study to assess the clinical, functional and radiological outcomes of the CE-marked ACE Acetabular Cup System. This is done by examining patient outcomes through questionnaires, reviews of X-rays and complications by patients who have received a total hip replacement using the ACE Acetabular Cup System at participating sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients deemed suitable for elective primary THR, as per indications in the IFU.
* Male or female, 18 years or older.

Exclusion Criteria:

* Patients who are unable to provide written informed consent.
* Patients deemed unsuitable for THR, as per contra-indications in the IFU.
* Patients indicated for THR as a result of trauma (i.e. neck of femur fracture).
* Patients who are pregnant (exclusion criteria for THR in general).
* Patients receiving implants other than the approved combination, i.e. an ACE Acetabular Cup System with a JRI femoral stem and head.
* Patients who are unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require elective primary total hip replacement
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
Oxford Hip Score | 3 years post-op
  A patient completed functional score to assess pain and function of the affected hip joint. Score range: 0 (worse) to 48 (best)

SECONDARY OUTCOMES:
Implant Survivorship | 6 months, 1 year, 3 years, 5 years, 7 years and 10 years post-op
  Implant survivorship based on revision rate and determined using the Kaplan-Meier analysis method
Oxford Hip Score | 6 months, 1 year, 5 years, 7 years and 10 years post-op
  A patient completed functional score to assess pain and function of the affected hip joint. Score range: 0 (worse) to 48 (best)
Modified Harris Hip Score | 6 months, 1 year, 3 years, 5 years, 7 years and 10 years post-op
  A patient completed functional score to assess pain and function of the affected hip joint. Score range: 0 (worse) to 100 (best)
EQ-5D-5L | 6 months, 1 year, 3 years, 5 years, 7 years and 10 years post-op
  A patient completed functional score to assess quality of life of the patient. Score range: -0.594 (worse) to 1.0 (best).
Radiological Assessment | 1 year, 5 years and 10 years post-op
  Radiographs reviewed for signs of radiolucencies, osteolysis, sclerosis and atrophy around the device

OTHER OUTCOMES:
Adverse Device Effects | 6 months, 1 year, 3 years, 5 years, 7 years and 10 years post-op
  Trends and anaylsis or adverse device effects reported

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Sussex NHS Foundation Trust, Worthing, United Kingdom

IPD SHARING:
Plan to Share IPD: No